CLINICAL TRIAL: NCT06648499
Title: Five Times Sit-To-Stand Test for Patients with Pediatric-Onset Multiple Sclerosis: Performance and Explanatory Factors
Brief Title: Five Times Sit-To-Stand Test for Patients with Pediatric-Onset Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yonca Zenginler Yazgan, Associate Professor, Istanbul University - Cerrahpasa
Other Study IDs: IUC-2024-152
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pediatric-Onset Multiple Sclerosis (POMS)
Keywords: lower extremity muscle strength; pediatric-onset multiple sclerosis; five times sit-to-stand test; physiotherapy
MeSH Terms: interventions — Exercise; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric-Onset Multiple Sclerosis Group: Individuals in the POMS group will be evaluated in terms of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue.
  Interventions: Other: Evaluation of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue in POMS
- Healthy Controls: Individuals in the control group will be evaluated in terms of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue.
  Interventions: Other: Evaluation of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue in healthy controls

INTERVENTIONS:
Other: Evaluation of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue in POMS — The demographic information of the patients will be taken with the form prepared for the people in this group. Patients will be assessed using the FTSTS test to evaluate lower extremity muscle strength, the Godin Leisure Time Exercise Questionnaire (GLTEQ) for physical activity, the 2-Minute Walk Test (2MWT) for exercise capacity, the Timed Up and Go (TUG) Test for functional mobility, the Pediatric Quality of Life Inventory (PedsQL) for quality of life, and the PedsQL Multidimensional Fatigue Scale for fatigue. All assessments will be completed on the same day and will not be repeated after a certain period of time.
  Groups: Pediatric-Onset Multiple Sclerosis Group
Other: Evaluation of lower extremity muscle strength, physical activity, exercise capacity, balance, quality of life, and fatigue in healthy controls — The demographic information of the healthy controls will be taken. Healthy controls will be assessed using the FTSTS test to evaluate lower extremity muscle strength, the Godin Leisure Time Exercise Questionnaire (GLTEQ) for physical activity, the 2-Minute Walk Test (2MWT) for exercise capacity, the Timed Up and Go (TUG) Test for functional mobility, the Pediatric Quality of Life Inventory (PedsQL) for quality of life, and the PedsQL Multidimensional Fatigue Scale for fatigue. All assessments will be completed on the same day and will not be repeated after a certain period of time.
  Groups: Healthy Controls

SUMMARY:
Transitioning from a sitting to a standing position is a movement essential for maintaining physical independence and functional mobility, and is necessary for performing many activities in daily life. Lower extremity muscle strength is considered the most critical factor reducing the capacity to perform the sit-to-stand movement. A study concluded that the Five-Times Sit-to-Stand test in patients with multiple sclerosis (MS) is multifactorial and is associated with walking speed and fatigue. Another study using the same test concluded that lower extremity capacity is reduced compared to healthy controls and is associated with balance, functional mobility, gait, and fatigue.

Pediatric-onset MS, occurring in patients under the age of 18, accounts for approximately 3-10% of all multiple sclerosis cases and is increasingly recognized in many parts of the world. According to our research, no studies have been found that demonstrate the extent of lower extremity involvement in patients with pediatric-onset MS compared to their healthy controls. Our aim is to evaluate the performance of the Five-Times Sit-to-Stand test in patients with pediatric-onset MS, compare it with healthy controls, and examine its relationship with physical activity, exercise capacity, functional mobility, quality of life and fatigue.

DETAILED DESCRIPTION:
In addition to visual, sensory, motor, and coordination impairments, cognitive problems, pain, and fatigue may occur in patients with pediatric-onset MS. Studies have reported that patients with pediatric-onset MS tend to participate in less physical activity and have lower exercise capacity compared to their healthy peers. Lower extremity functional capacity is impaired in most patients with MS, and the high prevalence of walking disorders is an example of this. Therefore, assessing lower extremity capacity and identifying modifiable determinants appears to be important. Moreover, a detailed assessment of lower extremity parameters in MS patients is crucial for determining appropriate rehabilitation programs. Transitioning from a sitting to a standing position is necessary for performing many activities in daily life. Assessment of lower extremity muscle strength using the sit-to-stand movement enables the development of preventive interventions in the early stages of the disease.

Our aim is to evaluate the performance of the Five-Times Sit-to-Stand (FTSTS) test in patients with pediatric-onset MS, compare it with healthy controls, and examine its relationship with physical activity, exercise capacity, functional mobility, quality of life, and fatigue. Under the supervision of a physical therapist, participants will be assessed using the FTSTS test to evaluate lower extremity muscle strength, the Godin Leisure Time Exercise Questionnaire (GLTEQ) for physical activity, the 2-Minute Walk Test (2MWT) for exercise capacity, the Timed Up and Go (TUG) Test for functional mobility, the Pediatric Quality of Life Inventory (PedsQL) for quality of life, and the PedsQL Multidimensional Fatigue Scale for fatigue.

It is planned to include 30 patients with pediatric-onset MS and 16 healthy controls, making a total of 46 participants in this study. The Shapiro-Wilk test will be employed to assess whether the data adhere to a normal distribution. Differences between groups will be analyzed using the independent sample t-test for normally distributed variables and the Mann-Whitney U test for non-normally distributed variables. The Chi-square test will be used to compare categorical variables. Intercorrelations among FTSTS and other variables will be calculated using Pearson or Spearman correlation analysis. This will be the first study to evaluate the performance of the FTSTS test in patients with pediatric-onset MS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate
* Being diagnosed with pediatric onset multiple sclerosis
* Being between the ages of 15-22
* EDSS ≤6

Exclusion Criteria:

* Having another diagnosis in addition to the diagnosis of pediatric-onset multiple sclerosis
* Having had an attack or received corticosteroid treatment 3 months before participating in the study

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample size was calculated based on the total fatigue scores in patients with pediatric-onset MS and healthy controls of the same age group, using the child form of the PedsQL Multidimensional Fatigue Scale as employed by Gravesande et al., with a 0.05 margin of error and 80% power. According to this calculation, it was seen that 25 patients with pediatric-onset MS and 13 healthy individuals who were matched for age and sex (2:1 distribution) should be included in our study. ). Considering the possibility of dropouts, we planned to include 30 patients with pediatric-onset MS and 16 healthy controls, making a total of 46 participants, with an additional 20% added to each group.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2024-11-18 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Five Times Sit-To-Stand Test performance | baseline
  The Five Times Sit-To-Stand Test is considered to be a valid, reliable, easy, and rapid method for evaluating lower extremity muscle strength in patients with MS. The time taken to complete five repetitions of the sit-to-stand movement will be measured as part of the test. Participants, seated in a chair without arm supports with their arms crossed over their chest, were instructed to stand up and sit down five times and to perform the test as quickly as possible. No encouragements will be given during the test. Prior to commencing, the participant will be instructed on how to perform the test, and an untimed practice trial will be conducted.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory | baseline
  Quality of life will be assessed using the Pediatric Quality of Life Inventory. This inventory contains two parallel forms, allowing both the child and the family to respond, and it is composed of sections on physical functioning, emotional functioning, social functioning, and school functioning. The total score is calculated on a scale from 0 to 100, with higher scores indicating better health-related quality of life.
PedsQL Multidimensional Fatigue Scale | baseline
  The fatigue levels of participants will be assessed using the PedsQL Multidimensional Fatigue Scale. The scale is a valid and reliable instrument for evaluating fatigue in pediatric populations. It consists of 18 items and covers 3 domains of fatigue (general, sleep/rest, and cognitive). Higher scores indicate greater levels of fatigue.
The Godin Leisure Time Exercise Questionnaire | baseline
  The Godin Leisure Time Exercise Questionnaire (GLTEQ) will be used to evaluate physical activity levels. GLTEQ is a self-reported questionnaire that is valid for PwPOMS measuring participants' physical activity behaviors. The first question inquires about the frequency of light, moderate, and vigorous physical activities that patients engage in for more than 15 minutes during a week. The second question of the survey asks about the frequency of activities performed in a week that are intense enough to induce sweating.
2-Minute Walk Test | baseline
  The 2-minute walk test (2MWT) is used to assess exercise capacity. The 2MWT has been reported to be a reliable and valid measure in PwMS. Participants will be instructed to cover as much distance as possible in 2 minutes on a 30-meter walking path in a single trial, and the total distance walked was recorded in meters.
Timed Up and Go Test | baseline
  The Timed Up and Go (TUG) test is an objective test used to assess functional mobility in patients with MS. In our study, prior to assessment, participants will be given an untimed trial to familiarize themselves with the test. Subsequently, the participant will be instructed to rise from the chair, walk 3 meters at a comfortable pace, and return to the chair to sit down again. The test will be administered twice, and the average of these trials will be considered for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Güler MD, Study Chair — Istanbul University - Cerrahpasa